CLINICAL TRIAL: NCT00583115
Title: A Phase II Study of Gleevec® (Imatinib Mesylate, NSC 716051 Formerly ST1571) in Children With Pulmonary Hypertension
Brief Title: Safety Study of Gleevec® in Children With Pulmonary Hypertension
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Unable to enroll subjects
Sponsor: Indiana University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 0702-21; Internally funded (Other: Indiana University)
Record Dates: First submitted 2007-12-20; First posted 2007-12-31 (Estimated); Results first posted 2015-10-29 (Estimated); Last update posted 2015-10-29 (Estimated); Status verified 2015-09

CONDITIONS: Pulmonary Hypertension
MeSH Terms: conditions — Hypertension, Pulmonary | interventions — Imatinib Mesylate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Gleevec (Experimental): Drug taken orally 260mg/M2/day once per day
  Interventions: Drug: Gleevec

INTERVENTIONS:
Drug: Gleevec — 260 mg/M2/day, given once daily by mouth
  Other Names: Imatinib Mesylate

SUMMARY:
The purpose of this study is to find out if the drug, Gleevec, is safe and effective in treating children with Pulmonary Hypertension.

DETAILED DESCRIPTION:
Idiopathic pulmonary artery hypertension (IPAH) is a rare but progressive disease in children and adults with a very high mortality from right heart failure. Platelet derived growth factor (PDGF) has been implicated in the pulmonary artery remodeling and vascular proliferation that is a pathologic hallmark of IPAH. Animal and clinical data support the hypothesis that activation of the PDGF receptor is critical in the development of IPAH, and inhibition of the PDGF signaling pathways may be a potential therapeutic target. Gleevec is a tyrosine kinase inhibitor developed for treatment of certain cancers and inhibits the PDGF receptor. Animal and preliminary clinical data suggest that Gleevec can reverse vascular remodeling and improve right heart failure. A small clinical trial for adults with IPAH is ongoing in Europe, but there are no trials in children where the disease has a worse prognosis. This project is a phase II, single dose pilot study to generate the hypothesis that activation of the PDGF receptor is critical in the development of IPAH, and inhibition of the PDGF signaling pathways is a potential therapeutic target. Five patients between the ages of 8 yr to 18 yr with severe IPAH will be recruited nationally, for a 6 month trial of Imatinib. The Specific Aim of this study is to collect preliminary data on the safety and efficacy of Gleevec in children with IPAH. Results from this study are needed to develop a larger, multi-center trial to determine the efficacy and therapeutic impact of Gleevec in children with IPAH. The long term goal of this work is to develop novel therapeutic strategies for treatment of IPAH in children. This translational study of the inhibition of the PDGF receptor in children with IPAH could provide insights into the etiology of IPAH and have a major impact on the development of new treatment strategies for both children and adults with pulmonary artery hypertension from multiple origins.

ELIGIBILITY:
Inclusion Criteria:

1. Male and female patients between the ages of 8 -18 years of age.
2. Diagnosis of idiopathic (or primary) pulmonary arterial hypertension according to the Venice Classification system (2003).54, 55
3. Functional classification of WHO class III - IV.
4. Pulmonary vascular resistance (PVR) >300 dynes / sec / cm5.
5. IPAH medications stable for at least 3 mo prior to baseline visit.
6. Female patients of child bearing potential who are sexually active must have negative pregnancy test within 7 days prior to initiation of study drug and use a double-barrier local contraception, i.e., intra-uterine device plus condom, or spermicidal gel plus condom up to the Study Completion visit.
7. Able to communicate well with the investigator, to understand and comply with the requirements of the study. Able to verbalize understanding and sign the written informed assent.
8. Parents, or legal guardians, must be able to communicate well with the investigator, to understand and comply with the requirements of the study. They must verbalize understanding and sign the written informed consent statement.

Exclusion Criteria:

1. Pre-existing lung disease including parasitic diseases affecting lungs, bronchial asthma, congenital abnormalities of the lungs, thorax and diaphragm.
2. Congenital heart disease, left ventricular failure, or left-sided obstructive lesion (pulmonary venous hypertension with pulmonary capillary wedge pressure > 12 mmHg) detected at right heart catheterization.
3. Chronic thromboembolic pulmonary hypertension, congenital or acquired deficiencies of blood coagulation, deficient thrombocyte function, thrombocytopenia < 40,000/μl, or Sickle Cell anemia.
4. Pregnancy, breast feeding, or lack of safe contraception (hormonal contraception, IUD, bilateral tubal ligation, hysterectomy) in premenopausal women.
5. Hepatic insufficiency with transaminase levels >4-fold the upper limit of normal, or a bilirubin > 2-fold the upper limit of normal.
6. Renal insufficiency (serum creatinine > 200 μmol/l).
7. History of clinically significant drug allergy or history of atopic allergy (asthma, urticaria, eczematous dermatitis). A known hypersensitivity to the study drug, or drugs similar to the study drug.
8. Previous therapeutic radiation of lungs or mediastinum.
9. Participation in any treatment studies within 3 months prior to dosing, or longer if required by local regulations, and for any other limitation of participation based on local regulations.
10. History of immunodeficiency diseases, including a positive HIV (ELISA and Western blot) test result, or a positive Hepatitis B surface antigen (HBsAg), or positive Hepatitis C test result.
11. Any surgical or medical condition which might significantly alter the absorption, distribution, metabolism or excretion of drugs, such as a history of inflammatory bowel syndrome, gastritis, ulcers, gastrointestinal or rectal bleeding, or a history of major gastrointestinal tract surgery such as gastrectomy, gastroenterostomy, or bowel resection.

    -

Ages: 8 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 1 (Actual)
Dates: Start 2007-10; Primary Completion 2013-08 (Actual); Study Completion 2013-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: R. Mark Payne, MD, Principal Investigator — Indiana University School of Medicine
Locations (1):
- Indiana University School of Medicine; Riley Hospital for Children, Indianapolis, Indiana, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Gleevec
Started | 1
Completed | 0
Not Completed | 1
Not completed — Death | 1

BASELINE CHARACTERISTICS:
Arm/Group | Gleevec
Number analyzed (Participants) | 1
Age, Customized [Number; unit: years]
  Age 8-18 years | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 1
Region of Enrollment [Number; unit: participants]
  United States | 1

OUTCOME MEASURES:

1. Primary Outcome: 1) Safety and Tolerability as Determined by Laboratory Evaluation, Physical Examination, Echocardiographic Analysis, and Adverse Events, and 2) Efficacy as Determined by an Increase in the Non-encouraged 6 Minute Walk Test From Baseline.
Time Frame: 6 months
Population: Unable to measure safety and tolerability as the participant died prior to study completion. Laboratory evaluations not able to be measured as participant died. Physical examination, Echocardiographic and adverse events not able to be measured as participant died Unable to measure 6 minute walk test as participant died prior to study completion.
Arm/Group | Gleevec
Number analyzed (Participants) | 0

2. Secondary Outcome: 1) Decrease in Pulmonary Artery Pressures and Vascular Resistance as Determined by Cardiac Catheterization, 2) Time to Clinical Worsening,3) Survival.
Time Frame: 6 months
Population: The only participant died prior to study completion. Unable to measure pulmonary artery pressure and vascular resistance as only participant died prior to study completion. Unable to measure time to clinical worsening as only participant died. Survival should be counted as 0.
Arm/Group | Gleevec
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Arm/Group | Gleevec
Serious Adverse Events (participants affected / at risk) | 1/1
Other Adverse Events (participants affected / at risk) | 0/1
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Gleevec (N=1)
Death (Cardiac disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No